CLINICAL TRIAL: NCT03193242
Title: eAMS: The Electronic Asthma Management System
Brief Title: The Electronic Asthma Management System
Acronym: eAMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-052A
Record Dates: First submitted 2017-05-09; First posted 2017-06-20 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Asthma; Asthma Action Plan
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Electronic Asthma Management System: eAMS Intervention
  eAMS consists of simple questionnaire completed either through an app on a patient's smartphone or tablet computer, a computerized clinical decision support system which then processes these data to produce a set of asthma care recommendations for the clinician, and a printable asthma action plan that is given to patients. eAMS will also provide access to a patient-oriented asthma management tool called Breathe.
  Interventions: Other: Electronic Asthma Management System: eAMS
- Control (No Intervention): Electronic Asthma Management System: eAMS - Control
  At control sites, eligible clinicians will be offered access to the web-based clinician-oriented asthma action plan (AAP) educational module produced by the Lung Association, copies of the Canadian Asthma Guidelines, and standard fillable paper-based AAPs (the eAMS will be offered after study end).

INTERVENTIONS:
Other: Electronic Asthma Management System: eAMS — Electronic Asthma Management System: eAMS Intervention
  eAMS consists of simple questionnaire completed either through an app on a patient's smartphone or tablet computer, a computerized clinical decision support system which then processes these data to produce a set of asthma care recommendations for the clinician, and a printable asthma action plan that is given to patients. eAMS will also provide access to a patient-oriented asthma management tool called Breathe.
  Arms: Intervention

SUMMARY:
This study is an extension of a pilot study in which investigators developed and tested a computerized tool to help physicians to determine if their patients' asthma is well controlled, advise them on medication changes required according to the current level of control, and automatically generate an electronic version of the AAP, all based on patient responses to a questionnaire completed by patients on a tablet computer. In this phase patients will have the ability to complete the questionnaire on their smartphones, through a pre-downloaded app and will have access to an electronic asthma self-management app.

DETAILED DESCRIPTION:
Asthma is a common and potentially fatal chronic disease. An asthma action plan (AAP) is a written plan produced by a physician for a patient with asthma, to provide education and guidelines for self-management of worsening asthma symptoms. Studies have shown that AAPs effectively improve asthma control, but physicians fail to provide AAPs due to lack of time and adequate skills. Physicians also often fail to determine if their patients have good asthma control, and to adjust medications in response to patients' control level.

In a pilot study investigators developed and tested a computerized tool to help physicians to determine if their patients' asthma is well controlled, advise them on medication changes required according to the current level of control, and automatically generate an electronic version of the AAP, all based on patient responses to a questionnaire completed by patients on a tablet computer. In the pilot, investigators found that the tablet computers add a level of complexity to clinic flow. In this study patients will have the ability to complete the questionnaire on their smartphones, through a pre-downloaded app. Patients will also have access to an electronic asthma self-management tool called Breathe through which they can view their AAP and other asthma educational information.

The investigators hope that this system will eliminate the barriers that physicians face in determining asthma control, adjusting medications, and delivering an AAP, and will increase the frequency with which physicians are able to achieve these goals in patients with asthma. The objectives of the study are to determine the impact of this system on asthma action plan delivery by primary care physicians, the frequency of checking control level, and the frequency and appropriateness of asthma medication changes (in accordance with control). The investigators will also attempt to determine the impact of the system on hospitalisations, emergency room (ER) visits, unscheduled visits to the doctor, total visits to the doctor, days off work or school, nocturnal asthma symptoms, daytime asthma symptoms, daytime rescue puffer use, and quality of life, and to measure physicians' perceptions of and satisfaction with the system.

ELIGIBILITY:
Inclusion Criteria:

* Eligible physicians will include all primary care physicians at the 4 sites.
* Eligible patients will include:

patients with asthma, as determined by a validated electronic chart record search algorithm for asthma; patients >/= 16 years of age.

Exclusion Criteria:

* Patients who received an AAP within the last 6 months (from their primary care physician, a respirologist, or any other source).
* Pregnant patients will be excluded given that conventional AAP recommendations may not be appropriate in this population.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Received AAP | 12 Months
  The study's primary outcome will be the proportion of patients currently on a controller medication who received an AAP in the intervention sites compared to the control sites, over 1 year (as determined through an electronic chart review).

SECONDARY OUTCOMES:
Documented Asthma Control | 12 months
  The proportion of eligible patients who had asthma control documented
Any Medication Change | 12 months
  The proportion of eligible patients who had a medication change made
Appropriate Medication Change | 12 months
  The proportion of eligible patients who had an appropriate medication change made (based on asthma control, where ascertainable)
Healthcare utilization rate | 12 months
  Secondary outcomes collected through patient questionnaire will measure healthcare utilization.
Quality of life | 12 months
  Secondary outcomes collected through patient questionnaires will measure quality of life.
Health Care Utilization | 12 months
  Health care utilization will also be validated through linkage with health administrative databases.
System Use | 12 months
  Quantitative assessment of system use
System usability | First 6 months of intervention
  Specific questionnaire to collect data on tool usability.
Tool learnability | First 6 months of intervention
  Focus group/interview to collect qualitative data on tool usability

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Wise Elephant Family Health Team, Brampton, Ontario
  - St. Michael's Hospital, Toronto, Ontario